CLINICAL TRIAL: NCT06578741
Title: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis Post-Approval Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA 24-01
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Aortic Aneurysm; Pararenal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Other): Treatment with GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device)
  Interventions: Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device)

INTERVENTIONS:
Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) — Treatment with the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) in patients with Pararenal Abdominal Aortic Aneurysms and Thoracoabdominal Aortic Aneurysms

SUMMARY:
This study aims to confirm that the benefit-risk assessment of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) remains positive in real-world use and to ensure the adequacy of the TAMBE Device training program.

DETAILED DESCRIPTION:
A maximum of 300 adult subjects will be enrolled at up to 60 U.S. centers, with a minimum of 70 subjects enrolled at study centers with no prior experience using the TAMBE Device. Subjects will have follow-up at 1 month, 6 months, 12 months and annually thereafter through 10 years post implant.

ELIGIBILITY:
Inclusion Criteria:

The subject is / has:

1. Treated with the aortic component of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Aortic Component) to allow endovascular repair of an aortic disease involving the visceral vessels.
2. Age ≥18 years at the time of informed consent signature.
3. An Informed Consent Form signed by subject or legal representative.

Exclusion Criteria:

The subject is / has:

1. Any contraindications for the TAMBE Device according to the IFU.
2. Planned parallel grafting with the TAMBE Aortic Component.
3. Intent to modify TAMBE Aortic Component (e.g., in situ fenestration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Co-Primary Endpoint #1: Technical Success | Time of index procedure
  All of the qualifying criteria are met (in the absence of surgical conversion or mortality, type I or type III endoleak, branch occlusion, or graft limb obstruction):
  * Successful access to the arterial system using remote arterial exposure, percutaneous technique, or open surgical conduits at index procedure.
  * Successful delivery and deployment of the aortic stent graft and all modular stent graft components at index procedure
  * Successful side branch catheterization and placement of bridging stents with restoration and maintenance of flow in all intended target vessels at final completion angiography.
  * Absence of type I or type III endoleaks at final completion angiography.
  * Patency of all aortic modular stent graft components and intended side branch components at final completion angiography.
Co-Primary Endpoint #2: Clinical Success | Index procedure through 12 months
  All of the following qualifying criteria are met from the initiation of the index procedure through 12 months post-index procedure:
  * Technical success
  * Absence of death from the initial procedure, secondary intervention, or aorta-related cause
  * Absence of persistent type I or type III endoleak
  * Absence of lesion enlargement >5 mm
  * Absence of device migration >10 mm
  * Absence of failure due to device integrity issues (defined as Grade 2 or 3 in Table 8)
  * Absence of lesion rupture
  * Absence of conversion to open surgical repair
  * Absence of permanent paraplegia (see definition below)
  * Absence of disabling stroke (see definition below)
  * Absence of "loss of function" or "end-stage renal disease" stage according to the RIFLE Classification following the index procedure

SECONDARY OUTCOMES:
Target Vessel Technical Success | 30 days, 6 months, annually through 10 years
  Successful catheterization and stent placement in all intended target vessels. Note: For this study, technical success will be reported for the overall procedure and specifically for the vessels targeted for treatment with the branch components (this "target vessel technical success" definition).
Secondary Clinical Success | 30 days, 6 months, annually through 10 years
  Initial clinical success that is interrupted by a treatment failure and is successfully corrected with secondary reintervention (e.g., a patient undergoes a successful treatment of a type I, II, or III endoleak).
Assisted Primary Clinical Success | 30 days, 6 months, annually through 10 years
  Clinical success that is obtained initially and continuously maintained with additional secondary reinterventions thus no interruption to initial clinical success.
Thirty-Day Mortality | 30 days
  Any death that occurs during the procedure, within the index procedure hospital stay, or within the first 30 days post-index procedure.
Lesion-Related Mortality | 30 days, 6 months, annually through 10 years
  Any death that occurs within the first 30 days, or any death that results from lesion rupture, aorta-related complications (e.g., infection, occlusion, dissection, hematoma), or a complication of a secondary intervention.
Major Adverse Events (MAEs) | 30 days, 6 months, annually through 10 years
  Includes any of the following:
  * All-cause mortality;
  * Myocardial infarction resulting in severe hemodynamic dysfunction necessitating resuscitation, cardiac arrest, or fatal outcome;
  * Respiratory failure requiring prolonged (>24 hours from anticipated) mechanical ventilation or reintubation;
  * Renal function decline characterized by one or more of the following:
    * >50% reduction in baseline Estimated Glomerular Filtration Rate (eGFR); or,
    * New-onset dialysis;
  * Bowel ischemia requiring surgical resection or not resolving with medical therapy;
  * Permanent paraplegia (see "permanent paraplegia" definition below)
  * Any major stroke
Secondary interventions | Time of index procedure
  Any Reintervention: Any repeated vascular or nonvascular procedure on the index device (TAMBE Device or any stent or stent graft in contact with any TAMBE component).
  • Note: Reintervention will be classified as "major", "minor", or "nonvascular" based on the definitions below.
  Major Reintervention: Deployment of proximal or distal extensions, removal of the device, use of thrombectomy or thrombolysis, and any major open surgical procedure.
  Minor Reintervention: Endovascular procedures (percutaneous transluminal angioplasty, atherectomy, stenting) without thrombectomy or thrombolysis, interventions to treat branch vessel stenosis, interventions to treat type II endoleaks or branch-related endoleaks, and minor surgical revisions (patch angioplasty) of the access vessels.
  Nonvascular Reinterventions: Any reinterventions that would not be considered "major reintervention" or "minor reintervention" based on the above definitions.
Intraprocedural Complications | 30 days, 6 months, annually through 10 years
  Any vessel perforation, dissection, or occlusion during target vessel cannulation and/or stenting.
Kink | 30 days, 6 months, annually through 10 years
  Objective documentation of demonstrable angulation (localized angle of less than 90 degrees when measured along the centerline) in any of the stent components or native target vessel
Stenosis | 30 days, 6 months, annually through 10 years
  Objective documentation of presence of narrowing with demonstrable flow in any of the components
Occlusion | 30 days, 6 months, annually through 10 years
  Objective documentation of presence of complete stent occlusion with or without minimal flow into a targeted vessel.
  Note: Occlusions will be stated if they occurred in the aortic component, in a branch component, or in a contralateral leg component used to treat the aortic disease.
Target Vessel Instability | 30 days, 6 months, annually through 10 years
  Any death or rupture related to side branch complication (e.g., endoleak) or any secondary intervention indicated to treat a branch-related complication, including endoleak, disconnection, kink, stenosis, occlusion, or rupture.
Secondary Patency | 30 days, 6 months, annually through 10 years
  Endovascular restoration of patency after occlusion of the side branch, stent, or stent graft has already occurred.
  Note: Conversion to bypass or inability to treat by endovascular means defines loss of secondary patency.
Primary Assisted Patency | 30 days, 6 months, annually through 10 years
  Endovascular intervention performed to maintain patency in the presence of stenosis before occlusion.
Primary Patency | 30 days, 6 months, annually through 10 years
  Uninterrupted patency with no occlusion or procedure performed to maintain patency on the stent or native target vessel.
  Note: Interventions intended to treat endoleak or stent disconnection do not count as loss of primary patency.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol